CLINICAL TRIAL: NCT04107415
Title: The Effect of Yoga on Respiratory Functions, Symptom Control and Life Quality of Asthma Patients: Randomized Controlled Study
Brief Title: The Effect of Yoga on Respiratory Functions, Symptom Control and Life Quality of Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, gülcan bahcecioğlu, Doctor Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-10/2
Record Dates: First submitted 2019-09-21; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Asthma; Yoga
Keywords: Asthma; nursing; patient; yoga
MeSH Terms: conditions — Asthma | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Randomization; participants were divided into two groups by using simple random numbers table, and then the first group which was drawn by lot method was named as the experimental group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga group (Experimental): group doing yoga
  Interventions: Other: yoga
- No yoga group (No Intervention): group not doing yoga

INTERVENTIONS:
Other: yoga — A total of 12 yoga sessions, 2 sessions a week for 6 weeks, was applied to the patients in the experimental group.
  Arms: Yoga group

SUMMARY:
This study was conducted to find out the effect of yoga applied to asthma patients on the patients' respiratory functions, symptom control and quality of life.

DETAILED DESCRIPTION:
While there are studies conducted with yoga on different patient groups in Turkey, no studies have been found on asthma patients specifically. For this reason, it was thought that studies are needed which will prove the effect of yoga practices in preventing and controlling symptoms of asthma patients and which will contribute to nursing literature.

ELIGIBILITY:
Inclusion Criteria:

* must be between 18 and 55 years old
* must be diagnosed with asthma at least for six months,
* must be living in the city centre,
* must be literate and volunteered to participated in the study, were included in the study

Exclusion Criteria:

* be participated in a regular exercise program in the last 6 months,
* be have another respiratory system disease
* be in the exacerbation period,
* have a physical disease or cognitive deficiency and a psychiatric disease diagnosis that could prevent understanding the training given,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Asthma Quality of Life Questionnaire | 6 week
  Performed to determine the quality of life of asthma patients. Asthma Quality of Life Questionnaire , which addresses both the physical and emotional aspects of the disease has 32 items and four sub-dimensions. These sub-dimensions are activity limitation (items 1, 2, 3, 4, 5, 11, 19, 25, 28, 31, 32), symptoms (items 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 29, 30), emotional functions (items 7, 13, 15, 21, 27) and environmental stimulants (items 9, 17, 23, 26). The scale is a 7-Likert type scale with "1" having the lowest point and "7" the highest point. Weights for the points of the questions are equal. General quality of life is calculated with the averages of all questions, while sub-dimensions are calculated by adding the scores of the related fields. Total score of the scale differs between 32 and 224. Higher total score and sub-dimension score averages mean higher quality of life. diagnosis
Asthma Control Test | 6 week
  The test consists of 5 questions. In this 5-Likert type scale, the scores of the answers are added up and the patient's state is evaluated. The maximum score one can get from this test is 25, while the minimum score is 5. While scoring Asthma Control Test, 25 points is accepted as "full control", 20-24 points is accepted as "good control" and less than 19 points is accepted as "no control". The highest score indicates the best control, while scores less than 19 indicate that the disease is not under control and that modifications should be made in the treatment to reach control.
Respiratory Function tests | 6 week
  Respiratory Function tests is a physiological parameter. Respiratory Function tests are assessed to find out the degree of airway constriction with spirometer and also to find out whether the disease is reversible and to make asthma diagnosis. Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), peak expiratory flow rate (PEF) and FEV1/FVC measurements were used to evaluate airway constriction

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan Bahçecioğlu Turan, Dr., Principal Investigator — Ataturk Üniversty
Locations (1):
- Atatürk university nursing faculty, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
after the article is published

REFERENCES:
- [Background] Kavak F, Ekinci M. The Effect of Yoga on Functional Recovery Level in Schizophrenic Patients. Arch Psychiatr Nurs. 2016 Dec;30(6):761-767. doi: 10.1016/j.apnu.2016.07.010. Epub 2016 Jul 30. PMID 27888972
- [Derived] Bahcecioglu Turan G, Tan M. The effect of yoga on respiratory functions, symptom control and life quality of asthma patients: A randomized controlled study. Complement Ther Clin Pract. 2020 Feb;38:101070. doi: 10.1016/j.ctcp.2019.101070. Epub 2019 Oct 28. PMID 31679902

DOCUMENTS (1):
  • Study Protocol (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT04107415/Prot_000.pdf